CLINICAL TRIAL: NCT00362778
Title: Intensive Insulin Therapy in Non-diabetic Patients With Acute Myocardial Infarction and Hyperglycaemia
Acronym: INSUCOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Xavier Bosch, Dr, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The INSUCOR study
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes; Hyperglycemia; Acute Myocardial Infarction
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin

ARMS (1):
- Serum saline (Sham Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — intravenous continuous insulin infusion for 48 hours

SUMMARY:
Hyperglycemia at admission has been associated with bad prognosis in patients with acute myocardial infarction (AMI). The clinical benefit of intensive treatment with insulin has been evaluated in diabetic patients admitted to intensive care units. The aim of our study was to assess the short-term effects and the safety of strict glycemic control in subjects with AMI and hyperglycemia without a previous history of diabetes.

DETAILED DESCRIPTION:
Twenty-eight non-previously diabetic patients admitted with AMI and hyperglycemia were randomized to two treatment arms, administered during the first 48 hours: the intensive group (n=13) received intravenous insulin with target glycemia levels of 80-110mg/dL, while the conventional group (n=15) received subcutaneous insulin only when glycemia was ³ 160mg/dL. High-sensitivity C-reactive protein (HS-CRP) was determined at 48 hours and before discharge and an oral glucose tolerance test (OGTT) was performed at 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of AMI, either with or without ST segment elevation
2. Presence of high blood glucose at admission with no previously known diabetes mellitus (DM)

Exclusion Criteria:

1. Age under 18 years old
2. History of DM
3. Presence of other cardiopathies (dilated cardiomyopathy, valvular or hypertrophic heart disease)
4. Unstable AMI patients (haemodynamic instability or arrhythmic disorders)
5. Platelet aggregation or coagulation disorders
6. Severe conditions with an estimated short (under 1 year) life expectancy
7. Participation in other trials
8. Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Glycemic control | first 48 hours

SECONDARY OUTCOMES:
High-sensitivity C-reactive protein levels | At 48 hours and aat hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bosch, Principal Investigator — Cardiology Department. Hospital Clínic i Universitari Barcelona